CLINICAL TRIAL: NCT05920161
Title: Neural Mechanisms of Stress Effects Across Hippocampal Encoding and Prediction
Brief Title: Influence of Stress on Encoding and Prediction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000030825; 1R21MH128740-01A1 (NIH)
Record Dates: First submitted 2023-06-15; First posted 2023-06-27 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Stress; Learning, Spatial
Keywords: memory
MeSH Terms: conditions — Spatial Learning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute Stress (Experimental): Participants complete the socially evaluated cold pressor test (SECPT), a validated laboratory-based stress induction procedure involving submerging an arm in an ice bath
  Interventions: Behavioral: Socially Evaluated Cold Pressor Test
- No Stress (Active Comparator): Participants complete a matched condition with no stress-related exposure involving submerging an arm in warm water
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Socially Evaluated Cold Pressor Test — The SECPT is a brief validated laboratory-based stress induction containing both physical and social elements
  Arms: Acute Stress
Behavioral: Control — This is matched to the SECPT but with warm instead of cold water
  Arms: No Stress

SUMMARY:
The purpose of this study is to investigate the neural mechanisms by which acute stress influences statistical learning and episodic encoding.

DETAILED DESCRIPTION:
This study aims to assess the neural and behavioral mechanisms by which acute stress modulates episodic encoding (which involves the trisynaptic pathway: entorhinal cortex, dentate gyrus, cornu ammonis [CA] 3, and CA 1) and statistical learning (monosynaptic pathway: entorhinal cortex, CA1) in humans.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old
* Fluent in English
* BMI 18-35

Exclusion Criteria:

* Meeting current DSM-V criteria for any substance use disorder (except caffeine)
* Having current significant medical conditions or psychiatric symptoms requiring medication
* Current use of medications/drugs that interfere with physiological stress responses
* Peri and post-menopausal women, pregnant or lactating women, and those with hysterectomies
* Metal in body (for MRI safety) history will be assessed for female participants.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth V Goldfarb, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate data will be shared on NIMH Data Archives

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 106 participants were randomized, 9 participants withdrew prior to receiving any intervention therefore 97 started
Period: Overall Study
Arm/Group | Acute Stress | No Stress
Started | 50 | 47
Analyzed for Behavior | 49 | 47
Analyzed for fMRI | 45 | 43
Completed | 50 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acute Stress | No Stress | Total
Number analyzed (Participants) | 49 | 47 | 96
Age, Continuous [Mean (Full Range); unit: years] | 23 [18 to 40] | 24 [18 to 45] | 24 [18 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 28 | 57
  Male | 20 | 19 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 45 | 41 | 86
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 17 | 20 | 37
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 20 | 17 | 37
  More than one race | 5 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 49 | 47 | 96

OUTCOME MEASURES:

1. Primary Outcome: Changes in fMRI Signal
Description: fMRI signal during learning will be assessed using connectivity, multivariate, and univariate approaches over 1-2 hour long learning period. Correlation between change in CA1-EC background connectivity and pair familiarity. rho represents the true correlation within the entire population, with values ranging from -1 to +1; values closer to +1 indicate a strong positive linear relationship, closer to -1 a strong negative one, and closer to 0 indicate no linear relationship.
Time Frame: 1-2 hours
Measure: Number; unit: Pearson's rho
Arm/Group | Acute Stress | No Stress
Number analyzed (Participants) | 45 | 43
Pearson's rho | 0.261 | -0.264
Statistical Analysis 1: Comparison: Acute Stress; Test type: Superiority; p = 0.023, t-test, 1 sided
Statistical Analysis 2: Comparison: No Stress; Test type: Superiority; p = 0.068, t-test, 1 sided

2. Primary Outcome: Statistical Learning
Description: Online measures of statistical learning ( mean reaction time) based on item predictability during task for condition A, B or x.
Time Frame: 1-2 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Acute Stress | No Stress
Number analyzed (Participants) | 49 | 47
minutes
  A condition | 0.692 (0.092) | 0.698 (0.078)
  B condition | 0.694 (0.094) | 0.694 (0.074)
  X condition | 0.686 (0.087) | 0.693 (0.070)
Statistical Analysis 1: Comparison: Acute Stress; Within-group A - B (null >0); Test type: Superiority; p = 0.281, t-test, 1 sided
Statistical Analysis 2: Comparison: No Stress; Within-group A - B (null >0); Test type: Superiority; p = 0.645, t-test, 1 sided
Statistical Analysis 3: Comparison: Acute Stress vs No Stress; Between-group comparison; Test type: Superiority; p = 0.245, t-test, 2 sided

3. Primary Outcome: Retention of Statistical Learning
Description: Offline measure of statistical learning assessed through familiarity tests the next day (comparison of accurate recognition of previously-studied pairs to chance, 50%)
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: correct pairs
Arm/Group | Acute Stress | No Stress
Number analyzed (Participants) | 49 | 47
correct pairs | 0.537 (0.247) | 0.477 (0.188)
Statistical Analysis 1: Comparison: Acute Stress; Test type: Superiority; p = 0.143, t-test, 1 sided
Statistical Analysis 2: Comparison: No Stress; Test type: Superiority; p = 0.797, t-test, 1 sided — above chance 0.5
Statistical Analysis 3: Comparison: Acute Stress vs No Stress; Test type: Superiority; p = 0.087, t-test, 2 sided

4. Primary Outcome: Episodic Memory
Description: Memory for individual items will be assessed through performance on old/new recognition tests the next day, quantified as hit rates and A' (non-parametric normalized ratio of hits to false alarms). Data presented here is the proportion of studied items attributed to the correct condition (A, B or X) minus the proportion of nonstudied items incorrectly attributed to that same condition.
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: proportion of items
Arm/Group | Acute Stress | No Stress
Number analyzed (Participants) | 49 | 47
proportion of items
  A condition | 0.067 (0.076) | 0.639 (0.072)
  B condition | 0.590 (0.079) | 0.619 (0.094)
  X condition | 0.615 (0.071) | 0.611 (0.073)
Statistical Analysis 1: Comparison: Acute Stress vs No Stress; A condition; Test type: Superiority; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Acute Stress vs No Stress; B condition; Test type: Superiority; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Acute Stress vs No Stress; X condition; Test type: Superiority; p < 0.0001, t-test, 2 sided

5. Secondary Outcome: Cortisol Reactivity
Description: Change in salivary cortisol levels following the SECPT/control procedure
Time Frame: 1-2 hours
Measure: Mean (Standard Deviation); unit: log nmol/L
Arm/Group | Acute Stress | No Stress
Number analyzed (Participants) | 49 | 47
log nmol/L | 0.636 (0.655) | -0.252 (0.475)
Statistical Analysis 1: Comparison: Acute Stress; Test type: Superiority; p < 0.000, t-test, 1 sided
Statistical Analysis 2: Comparison: No Stress; Test type: Superiority; p = 0.0008, t-test, 1 sided

6. Secondary Outcome: Alpha-amylase Reactivity
Description: Change in salivary alpha-amylase levels following the SECPT/control procedure
Time Frame: 1-2 hours
Measure: Mean (Standard Deviation); unit: log nmol/L
Arm/Group | Acute Stress | No Stress
Number analyzed (Participants) | 49 | 47
log nmol/L | -0.286 (1.270) | -0.281 (1.199)
Statistical Analysis 1: Comparison: Acute Stress; Test type: Superiority; p = 0.083, t-test, 1 sided
Statistical Analysis 2: Comparison: No Stress; Test type: Superiority; p = 0.088, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 2 days
Arm/Group | Acute Stress | No Stress
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/47
Other Adverse Events (participants affected / at risk) | 0/50 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT05920161/Prot_SAP_000.pdf
  • Informed Consent Form (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT05920161/ICF_001.pdf